CLINICAL TRIAL: NCT00751868
Title: NEO-ADIXERN (NEO-ADjuvant IXabepilone in Breast Cancer). A Feasibility Study of Dose-dense FEC With G-CSF Support Followed by Dose-dense Ixabepilone With G-CSF Support as Neoadjuvant Chemotherapy in Breast Cancer
Brief Title: FEC With G-CSF Support Followed by Ixabepilone With G-CSF Support as Neoadjuvant Chemotherapy in BC
Acronym: GIM9
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Consorzio Oncotech (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIM9-NEO-ADIXERN
Record Dates: First submitted 2008-09-11; First posted 2008-09-12 (Estimated); Last update posted 2014-12-17 (Estimated); Status verified 2014-12

CONDITIONS: Breast Cancer
Keywords: breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — ixabepilone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ARM 1 (Experimental): FEC e Ixabepilone. A goal of 48 patients will be enrolled in this study by 16 Italian centres of the GIM (Gruppo Italiano Mammella) Group. Subjects must meet all of the inclusion criteria and none of the exclusion criteria to be enrolled in the study
  Interventions: Drug: Ixabepilone

INTERVENTIONS:
Drug: Ixabepilone — Ixabepilone is administered as 3-hour intravenous infusion (iv) at the dose of 40 mg/mq, every 14 days for 4 cycles (with G-CSF support), sequentially to Fluorouracil 600 mg/mq as intravenous (iv) infusion, Epirubicin 90 mg/mq as intravenous (iv) bolus and Cyclophosphamide 600 mg/mq as intravenous (iv) infusion every 14 days for 4 cycles (with G-CSF support)
  Other Names: Ixempra

SUMMARY:
The purpose of this study is to assess the feasibility of Ixabepilone (4 cycles) administered every 14 days with the support of G-CSF sequentially to the combination of Fluorouracil, Epirubicin and Cyclophosphamide (4 cycles) administered every 14 days with the support of G-CSF.

To evaluate the efficacy (in terms of pathologic Complete Responses in the breast and in the axilla), the dose reduction rate, the median treatment delay and the discontinuation rate due to toxicity of the regimen.

DETAILED DESCRIPTION:
Estrogen receptor negative breast cancer may be defined as distinct biologic subtype disease, more aggressive with a typical molecular portrait. [30] This subtype seems to have a poor prognosis and poor treatment options because these patients are not candidate to hormonal therapy. Novel treatment strategies focusing upon this subtype are necessary in the future. [31] There are reports of clinical benefit in estrogen receptor negative patients treated with dose-dense chemotherapy (see background CALGB 9741 and MIG-1 study). In the CALGB 9741 study, patients randomized to receive dose-dense regimens experienced severe toxicities during paclitaxel treatment leading to dose reduction in 7% and 5%respectively.

Ixabepilone has shown consistent activity and an acceptable safety profile in patients with all stages breast cancer. This phase II study evaluate the feasibility of dose-dense Ixabepilone (4 cycles) given sequentially to the combination of Fluorouracil, Epirubicin and Cyclophosphamide (4 cycles) all given every 14 days with the support of Filgrastim as neo-adjuvant treatment for ER-negative breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Histological documented diagnosis of breast cancer by incisional biopsy
* Clinical T>=2
* Females age >= 18 and <= 70 years
* ECOG performance status 0-1
* No prior treatment for breast cancer excluding therapy for DCIS
* Subjects with hormone replacement therapy are eligible if this therapy is discontinued at least 2 weeks before starting therapy
* Neutrophils > 2x109/L, Hgb > 9 g/dL, platelets > 100x109/L
* Total bilirubin < 1 time the upper limit of normal (ULN) of the Institutional normal values and AST and/or ALT < 2.5 ULN, alkaline phosphatase < 2.5 ULN
* Serum creatinine < 1.5 times the upper limit of normal (ULN)
* Normal cardiac function (normal ECG required in all patients, normal ECG and MUGA or Echocardiography with EF only in HER-2 positive patients)
* Negative pregnancy test prior to inclusion in the study (if potentially childbearing)
* Signed Informed consent

Exclusion Criteria:

* Prior or current history of ipsilateral or controlateral breast invasive cancer. A past or current history of ipsilateral ductal carcinoma in situ or ipsilateral/controlateral lobular neoplasia in situ are not an exclusion criteria as well as a controlateral ductal carcinoma in situ removed by mastectomy
* Inflammatory breast cancer
* Metastatic breast cancer (M1)
* Histology other than adenocarcinoma of the breast
* Male patients
* Pregnant or lactating women or women of childbearing potential (e.g. not using adequate contraception)
* Patients unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for up to 8 weeks after the last dose of investigational drug
* History of prior or concomitant malignancies other than curatively treated basal cell skin cancer or excised cervical carcinoma in situ
* Symptomatic peripheral neuropathy > grade 1 according to the NCI CTC
* Other serious illness or medical condition:
* Congestive hearth failure or angina pectoris even if it is medically controlled. In particular, Ejection Fraction (EF) below the Institutional normal value for MUGA Fraction (EF) below the Institutional normal value for MUGA, or below 50% for ECHO
* Previous history of myocardial infarction uncontrolled, high-risk ipertension or arrhythmia
* History of significant neurological or psychiatric disorders including dementia or seizures
* Active infection, active peptic ulcer, unstable diabetes mellitus or contraindications for the use of steroids
* History of previous or concomitant malignancies other than curatively treated basal cell skin cancer or excised cervical carcinoma in situ
* Concurrent treatment with other experimental drugs. Participation in another clinical trial with any investigational regimen within 30 days prior to study entry
* Prior severe HSR to agents containing Cremophor EL

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2008-09; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Pathologic Complete Response (pCR) | one year

SECONDARY OUTCOMES:
Feasibility/Tolerability for an individual patient is defined as the absence of hematologic toxicities requiring dose reduction as per protocol | one year

CONTACTS AND LOCATIONS:
Overall Officials: Marco MV Venturini, Doctor, Principal Investigator — Ospedale Sacro Cuore - Dipartimento di Oncologia Medica
Locations (15):
- Italy (15):
  - Azienza Osped.Treviglio - Caravaggio, Treviglio, BG
  - Azienda Ospedaliera G. Rummo, Benevento, BN
  - Ospedale Civile di Campobasso - A. Cardarelli, Campabasso, CB
  - Ospedale civile Renzetti di Lanciano, Lanciano, CH
  - Azienda Ospedaliera S. Anna, Como, CO
  - Azienda Ospedaliera Nesina Garibaldi, Catania, CT
  - I.S.T. - Istituto Nazionale per la Ricerca sul Cancro, Genova, GE
  - Presidio Ospedaliero di Macerata, Mecerata, MC
  - I.R.C.C.S. Multimedica - Casa di Cura Accreditata, Sesto San Giovanni, Milano
  - Azienda Ospedaliera R. Silvestrini, Perugia, PG
  - Istituto Regina Elena, Roma, Roma
  - Azienda Ospedaliera SS. Annunziata, Sassari, SS
  - Ospedale S. Cuore Don Calabria, Negrar, Verona
  - Ist. Nazionale per lo Studio e la Cura dei Tumori - Fondazione Pascale, Napoli
  - Università Federico II, Napoli

REFERENCES:
- [Derived] Clavarezza M, Bordonaro R, Daniele B, Ferrandina G, Barni S, Turazza M, Coati F, De Matteis A, De Placido S, Cognetti F, Olmeo NA, Carrozza F, Bruzzi P, Del Mastro L; Gruppo Italiano Mammella. Dose-dense FEC followed by dose-dense ixabepilone as neoadjuvant treatment for breast cancer patients: a feasibility study. Oncologist. 2013;18(8):924-5. doi: 10.1634/theoncologist.2013-0222. Epub 2013 Aug 12. PMID 23939283